CLINICAL TRIAL: NCT00374322
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled Study of Adjuvant Lapatinib (GW572016) in Women With Early-Stage ErbB2 Overexpressing Breast Cancer
Brief Title: Tykerb Evaluation After Chemotherapy (TEACH): Lapatinib Versus Placebo In Women With Early-Stage Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EGF105485
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-07

CONDITIONS: Neoplasms, Breast
Keywords: Breast Cancer; ErbB2-overexpressing; early-stage breast cancer; adjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 6 tablets daily for 12 months
  Interventions: Other: placebo
- Lapatinib (Experimental): Lapatinib 1500 mg (6 tablets) daily for 12 months
  Interventions: Drug: lapatinib

INTERVENTIONS:
Drug: lapatinib — Lapatinib 1500 mg (6 tablets) daily for 12 months
  Arms: Lapatinib
Other: placebo — 6 tablets daily for 12 months
  Arms: Placebo

SUMMARY:
This study was designed to evaluate and compare the safety and efficacy of an oral dual tyrosine kinase inhibitor, lapatinib, versus placebo in women with early-stage ErbB2-overexpressing breast cancer who have completed their primary neoadjuvant or adjuvant chemotherapy and have no clinical or radiographic evidence of disease.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed ErbB2-overexpressing invasive carcinoma (TX or T1-4) of the breast at the time of the initial diagnosis and have undergone adequate excision of tumor;
* Had tumors that overexpress ErbB2 defined as 3+ by IHC or c-erbB2 gene amplification by FISH (ErbB2 expression/amplification must be documented prior to study entry; however, a tumor tissue sample must be sent to a central laboratory for subsequent re-analysis of ErbB2 status);
* Have Stage I through Stage IIIc disease according to the American Joint Committee on Cancer (6th edition) staging criteria for breast cancer and meet one of the following criteria:

node-positive disease defined as: one positive lymph node by sentinel node biopsy OR at least 1 positive lymph node found among at least 6 axillary nodes examined on axillary node dissection OR status post axillary radiotherapy for sterilization if clinically evaluated as cN1 or cN2 (if sentinel node biopsy is positive, subject may either undergo an axillary node dissection or radiotherapy to the axilla).

node-positive disease evaluated as: ipsilateral axillary lymph nodes cN0-2 by clinical evaluation and axillary lymph nodes pNX, pN0(i+), or pN1-3 by pathological evaluation [patients with pN3 (Stage IIIc disease) must be disease free following completion of neoadjuvant or adjuvant chemotherapy for at least 12 months and must not have been lost to follow up].

OR node-negative disease defined as: negative sentinel node biopsy OR no positive lymph nodes found among at least 6 axillary nodes examined on axillary node dissection OR status post axillary radiotherapy for sterilization if clinically evaluated as cN0.

node-negative disease categorized as: high-risk disease (tumor >2.0 cm if ER and/or progesterone receptor (PgR) positive disease is present or tumor >1.0 cm if ER and PgR negative disease) OR intermediate-risk disease (tumor 1.0-2.0 cm and ER and/or PgR positive disease).

* Women with synchronous bilateral invasive breast cancer or synchronous DCIS of either the contralateral or ipsilateral breast at the time of the initial diagnosis are also eligible;
* Have undergone either mastectomy OR lumpectomy;
* Have received and completed treatment with a neoadjuvant or adjuvant chemotherapy regimen containing either an anthracycline or a taxane; or any cyclophosphamide, methotrexate and 5-fluorouracil (CMF) regimen;
* May continue to receive endocrine therapy while taking study medication, if endocrine therapy was initiated as either adjuvant therapy for treatment of the initial diagnosis of invasive breast cancer or for ovarian function suppression; however, endocrine therapy may not be initiated while taking study medication. Endocrine therapy agents may be switched while participating in this study (e.g., stop tamoxifen and start letrozole);
* May have received prior radiotherapy as treatment for primary tumor; however, is not required for study entry;
* May continue to receive radiotherapy while taking study medication, if radiotherapy was initiated as adjuvant therapy for treatment of the initial diagnosis of invasive breast cancer;
* May continue to receive bisphosphonates only for treatment of documented osteoporosis, but not as treatment or prophylaxis of bone metastases;
* All women eligible for adjuvant treatment with trastuzumab, including those diagnosed and treated within the last six months, must be considered for such treatment prior to being offered participation in this study. Participation in this study will be allowed only if the physician and patient have considered and discussed at length the advantages of trastuzumab, but have mutually decided against initiating trastuzumab therapy.
* Have clinical and radiologic assessments that are negative for local or regional recurrence of disease or metastatic disease at the time of study entry;
* if signs or symptoms suggestive of either recurrence of disease or metastatic disease are present, the appropriate radiological imaging must be performed
* if the following laboratory results are present, the appropriate radiological imaging must be performed:
* for AST/ALT ≥2×ULN or ALP ≥2×ULN (not in the bone fraction), an abdominal CT or MRI must be done
* for ALP≥2×ULN in the bone fraction, a bone scan must be done; a confirmatory x-ray, CT scan or MRI scan or biopsy is required if the results of the bone scan are inconclusive
* Have a unilateral/bilateral mammogram within 12 months prior to study entry;
* Have an analysis of both ER and PgR on the primary tumor prior to study entry;
* Have a cardiac ejection fraction within institutional range of normal as measured by either echocardiogram or multigated acquisition scans;
* Have an Eastern Cooperative Oncology Group Performance Status of 0 to 1;
* Women with a history of non-breast malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence. Women with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical carcinoma in situ, melanoma in situ, and basal cell or squamous cell carcinoma of the skin;
* Are able to swallow and retain oral medication;
* Have a paraffin-embedded tissue block from an archived tumor tissue from the primary tumor or twenty (20) slides of paraffin-embedded tissue available for biomarker analysis;
* Have adequate organ function defined as: absolute neutrophil count ≥1.5× 10^9/L; hemoglobin ≥9 g/dL; platelets ≥75 × 10^9/L; albumin ≥2.5 g/dL; serum bilirubin ≤1.25 ×ULN; aspartate aminotransferase and alanine aminotransferase ≤3 × ULN and serum creatinine ≤2.0 mg/dL or calculated creatinine clearance ≥40 mL/min
* Have signed the informed consent form (ICF);
* Women of child-bearing potential must have a negative serum pregnancy test at screening and agree to complete abstinence from intercourse or consistent and correct use of an acceptable methods of birth control from 2 weeks prior to administration of the first dose of study medication until 28 days after the final dose of study medication:

Exclusion Criteria:

* Have clinical and radiologic evidence of local or regional recurrence of disease or metastatic disease at the time of study entry;
* Had metachronous invasive breast cancer (breast cancers diagnosed at different times);
* Have a prior history of other breast cancer malignancies, including DCIS;
* Are unable to provide archived tumor tissue samples for assay;
* Had prior therapy with an ErbB1 and/or ErbB2 inhibitor; women who experienced a hypersensitivity or allergic reaction to trastuzumab during the first infusion and were unable to complete this infusion are eligible;
* Receive concurrent anti-cancer therapy (chemotherapy, immunotherapy, and biologic therapy) while taking study medication;
* Have unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior cancer treatment;
* Have malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Women with ulcerative colitis are also excluded;
* Have a concurrent disease or condition that would make the woman inappropriate for study participation, or any serious medical disorder that would interfere with the woman's safety;
* Have an active or uncontrolled infection;
* Have dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent;
* Have a known history of uncontrolled or symptomatic angina, arrhythmias, or CHF;
* Are pregnant or breastfeeding;
* Receive concurrent treatment with an investigational agent; women, who are in follow-up in another clinical trial where the primary endpoint has been met and the interval between assessments is ≥12 months and radiological imaging is not required at these assessments, are eligible;
* Receive concurrent treatment with a selected list of strong inducers and inhibitors of CYP3A4;
* Used an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study medication;
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to lapatinib or excipients;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3166 (Actual)
Dates: Start 2006-08; Primary Completion 2011-09 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (378):
- United States (94):
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Sedona, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Gilroy, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, La Verne, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fairfield, Connecticut
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Torrington, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Port Saint Lucie, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Joliet, Illinois
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Ames, Iowa
  - GSK Investigational Site, Sioux City, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Marrero, Louisiana
  - GSK Investigational Site, Scarborough, Maine
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Danvers, Massachusetts
  - GSK Investigational Site, Newton, Massachusetts
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Duluth, Minnesota
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Robbinsdale, Minnesota
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Saint Joseph, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Hooksett, New Hampshire
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Paramus, New Jersey
  - GSK Investigational Site, Sparta, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, East Setauket, New York
  - GSK Investigational Site, Mount Kisco, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Charleston, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Middletown, Ohio
  - GSK Investigational Site, Drexel Hill, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Duncanville, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Round Rock, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Chesapeake, Virginia
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Richlands, Virginia
  - GSK Investigational Site, Kirkland, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Vancouver, Washington
  - GSK Investigational Site, Yakima, Washington
- Argentina (9):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Neuquén, Neuquén Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Santa Fe, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Quilmes
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (22):
  - GSK Investigational Site, Campbelltown, New South Wales
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Kogarah, New South Wales
  - GSK Investigational Site, Liverpool, New South Wales
  - GSK Investigational Site, North Sydney, New South Wales
  - GSK Investigational Site, Douglas, Queensland
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Redcliffe, Queensland
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Elizabeth Vale, South Australia
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, East Melbourne, Victoria
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Footscray, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Parkville, Victoria
  - GSK Investigational Site, Ringwood East, Victoria
  - GSK Investigational Site, Wodonga, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
  - GSK Investigational Site, Perth, Western Australia
- GSK Investigational Site, Brussels, Belgium
- Brazil (5):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Rio de Janeiro, Rio de Janeiro
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Santo André, São Paulo
  - GSK Investigational Site, São Paulo, São Paulo
- Canada (14):
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan
- Chile (2):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- China (6):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
- Croatia (5):
  - GSK Investigational Site, Osijek
  - GSK Investigational Site, Pula
  - GSK Investigational Site, Rijeka
  - GSK Investigational Site, Split
  - GSK Investigational Site, Zagreb
- Czechia (2):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Prague
- Denmark (8):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Esbjerg
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Næstved
  - GSK Investigational Site, Odense
  - GSK Investigational Site, Roskilde
  - GSK Investigational Site, Vejle
- France (25):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Colmar
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montbéliard
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Saint-Cloud
  - GSK Investigational Site, Saint-Grégoire
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tourcoing
  - GSK Investigational Site, Vandœuvre-lès-Nancy
  - GSK Investigational Site, Villejuif
- Germany (77):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Konstanz, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Mayen, Baden-Wurttemberg
  - GSK Investigational Site, Mutlangen, Baden-Wurttemberg
  - GSK Investigational Site, Rheinfelden, Baden-Wurttemberg
  - GSK Investigational Site, Schwetzingen, Baden-Wurttemberg
  - GSK Investigational Site, Singen, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Amberg, Bavaria
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Bayreuth, Bavaria
  - GSK Investigational Site, Deggendorf, Bavaria
  - GSK Investigational Site, Ebersberg, Bavaria
  - GSK Investigational Site, Eggenfelden, Bavaria
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Fürth, Bavaria
  - GSK Investigational Site, Kempten (Allgäu), Bavaria
  - GSK Investigational Site, Krumbach, Bavaria
  - GSK Investigational Site, Marktredwitz, Bavaria
  - GSK Investigational Site, Memmingen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Rehling, Bavaria
  - GSK Investigational Site, Rosenheim, Bavaria
  - GSK Investigational Site, Roth, Bavaria
  - GSK Investigational Site, Schwandorf in Bayern, Bavaria
  - GSK Investigational Site, Weiden, Bavaria
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Fürstenwalde, Brandenburg
  - GSK Investigational Site, Bremen, City state Bremen
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Goslar, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Hildesheim, Lower Saxony
  - GSK Investigational Site, Salzgitter, Lower Saxony
  - GSK Investigational Site, Güstrow, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Herne, North Rhine-Westphalia
  - GSK Investigational Site, Hilden, North Rhine-Westphalia
  - GSK Investigational Site, Mülheim, North Rhine-Westphalia
  - GSK Investigational Site, Porta Westfalica, North Rhine-Westphalia
  - GSK Investigational Site, Recklinghausen, North Rhine-Westphalia
  - GSK Investigational Site, Troisdorf, North Rhine-Westphalia
  - GSK Investigational Site, Velbert, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Homburg/Saar, Saarland
  - GSK Investigational Site, Neunkirchen, Saarland
  - GSK Investigational Site, Saarbrücken, Saarland
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Kauschwitz, Saxony
  - GSK Investigational Site, Neustadt, Saxony
  - GSK Investigational Site, Spremberg, Saxony
  - GSK Investigational Site, Zittau, Saxony
  - GSK Investigational Site, Zwickau, Saxony
  - GSK Investigational Site, Blankenburg, Saxony-Anhalt
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Stendal, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Eisenach, Thuringia
  - GSK Investigational Site, Jena, Thuringia
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Chania
  - GSK Investigational Site, Heraklion, Crete
- Hong Kong (3):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Shatin
  - GSK Investigational Site, Wan Chai
- Hungary (6):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Kaposvár
  - GSK Investigational Site, Kistarcsa
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Szeged
- India (6):
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
- Israel (7):
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Tel Aviv
- Italy (6):
  - GSK Investigational Site, Avellino, Campania
  - GSK Investigational Site, Piacenza, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Perugia, Umbria
  - GSK Investigational Site, Negrar (Verona), Veneto
- Latvia (2):
  - GSK Investigational Site, Liepāja
  - GSK Investigational Site, Riga
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Klaipėda
  - GSK Investigational Site, Vilnius
- Mexico (5):
  - GSK Investigational Site, Chihuahua City, Chihuahua
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, DF.
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México D.F.
- New Zealand (3):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Hamilton
- GSK Investigational Site, Lima, Lima Province, Peru
- Philippines (4):
  - GSK Investigational Site, Baguio City, Benguet
  - GSK Investigational Site, Cebu
  - GSK Investigational Site, Pasig
  - GSK Investigational Site, Quezon City
- Poland (5):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Yaroslavl
- Slovakia (4):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Bardejov
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Nitra
- South Africa (9):
  - GSK Investigational Site, Tygerberg, Western Province
  - GSK Investigational Site, Athlone Park, Amanzimtoti
  - GSK Investigational Site, Groenkloof
  - GSK Investigational Site, Kraaifontein
  - GSK Investigational Site, Overport
  - GSK Investigational Site, Parktown
  - GSK Investigational Site, Port Elizabeth
  - GSK Investigational Site, Sandton
  - GSK Investigational Site, Saxonwold, Johannesburg
- South Korea (3):
  - GSK Investigational Site, Goyang-si, Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Songpa-gu, Seoul
- Spain (16):
  - GSK Investigational Site, Alcorcón
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Jaén
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Llobregat
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Ourense
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Santa Cruz de Tenerife
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- Ukraine (4):
  - GSK Investigational Site, Dnipro
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Uzhhorod
- United Kingdom (14):
  - GSK Investigational Site, Chelmsford, Essex
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Sutton, Surrey
  - GSK Investigational Site, Bournemouth
  - GSK Investigational Site, Edgbaston, Birmingham
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Lindley
  - GSK Investigational Site, London
  - GSK Investigational Site, Maidstone
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, Shrewsbury

REFERENCES:
- [Background] P Goss, I Smith, J O'Shaughnessy, B Ejlertsen, M Kaufmann, F Boyle, A Buzdar, P Fumoleau, W Gradishar, M Martin, B Moy, M Piccart-Gebhart, K I Pritchard, D Lindquist, Y Chavarri-Guerra, G Aktan, E Rappold, L S Williams, D M Finkelstein. Resubmission: A Randomized Trial of Adjuvant Lapatinib in Women with Early Stage HER2 Overexpressing Breast Cancer. Lancet Oncol. 2012;S 1470-2045(12):70508-9.
- [Derived] Boyle FM, Smith IE, O'Shaughnessy J, Ejlertsen B, Buzdar AU, Fumoleau P, Gradishar W, Martin M, Moy B, Piccart-Gebhart M, Pritchard KI, Lindquist D, Amonkar M, Huang Y, Rappold E, Williams LS, Wang-Silvanto J, Kaneko T, Finkelstein DM, Goss PE; TEACH Investigators. Health related quality of life of women in TEACH, a randomised placebo controlled adjuvant trial of lapatinib in early stage Human Epidermal Growth Factor Receptor (HER2) overexpressing breast cancer. Eur J Cancer. 2015 Apr;51(6):685-96. doi: 10.1016/j.ejca.2015.02.005. Epub 2015 Mar 6. PMID 25752740
- [Derived] Schaid DJ, Spraggs CF, McDonnell SK, Parham LR, Cox CJ, Ejlertsen B, Finkelstein DM, Rappold E, Curran J, Cardon LR, Goss PE. Prospective validation of HLA-DRB1*07:01 allele carriage as a predictive risk factor for lapatinib-induced liver injury. J Clin Oncol. 2014 Aug 1;32(22):2296-303. doi: 10.1200/JCO.2013.52.9867. Epub 2014 Mar 31. PMID 24687830
- [Derived] Goss PE, Smith IE, O'Shaughnessy J, Ejlertsen B, Kaufmann M, Boyle F, Buzdar AU, Fumoleau P, Gradishar W, Martin M, Moy B, Piccart-Gebhart M, Pritchard KI, Lindquist D, Chavarri-Guerra Y, Aktan G, Rappold E, Williams LS, Finkelstein DM; TEACH investigators. Adjuvant lapatinib for women with early-stage HER2-positive breast cancer: a randomised, controlled, phase 3 trial. Lancet Oncol. 2013 Jan;14(1):88-96. doi: 10.1016/S1470-2045(12)70508-9. Epub 2012 Dec 10. PMID 23234763

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women with early-stage ErbB2-overexpressing breast cancer who had not been previously treated with trastuzumab were enrolled in this Phase III study. Women who subsequently had no clinical or radiologic evidence of disease were enrolled after completion of primary neoadjuvant/adjuvant chemotherapy.
Pre-assignment Details: The study consisted of a Screening Period, a 1-year Treatment Period, and a Follow-up (FU) Period of up to 5 years after the date of study drug withdrawal/completion, for disease status/survival. A total of 3161 eligible participants (par.) (of the 3166 enrolled) were randomized, out of which 3147 par. received at least one dose of study treatment.
Groups:
- Lapatinib 1500 mg: Participants received lapatinib 1500 milligrams (mg) orally once daily. Treatment was continued for a maximum of 12 months or until disease recurrence or development of a second primary cancer, withdrawal from study treatment due to unacceptable toxicity, or consent withdrawal.
- Placebo: Participants received matching placebo orally once daily. Treatment was continued for a maximum of 12 months or until disease recurrence or development of a second primary cancer, withdrawal from study treatment due to unacceptable toxicity, or consent withdrawal.
Period: Overall Study
Arm/Group | Lapatinib 1500 mg | Placebo
Started | 1579 | 1582
Received >=1 Dose of Study Treatment | 1571 | 1576
Completed | 322 | 278
Not Completed | 1257 | 1304
Not completed — Lost to Follow-up | 92 | 90
Not completed — Protocol Violation | 8 | 3
Not completed — Withdrawal by Subject | 235 | 167
Not completed — Sponsor Terminated Study | 866 | 990
Not completed — Physician Decision | 36 | 32
Not completed — Par. Consented to Survival FU Only | 3 | 1
Not completed — Sponsor Decision | 2 | 3
Not completed — FU by a Non-Principal Investigator (PI) | 2 | 3
Not completed — Seen in FU by a Non-Primary Investigator | 1 | 0
Not completed — Severe Toxicity | 1 | 0
Not completed — Site Closed | 2 | 2
Not completed — Participant Changed Physician | 1 | 0
Not completed — Started Another Chemotherapy Regimen | 0 | 1
Not completed — Noncompliance with Study Requirements | 0 | 1
Not completed — Withdrew Consent During Follow-up | 0 | 5
Not completed — Did Not Receive Study Medication | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lapatinib 1500 mg | Placebo | Total
Number analyzed (Participants) | 1571 | 1576 | 3147
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.7 (9.89) | 52.3 (9.94) | 52.0 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1571 | 1576 | 3147
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Participants can appear in more than one race category.
  Participants
    African American/ African Heritage | 53 | 62 | 115
    American Indian or Alaskan Native | 65 | 67 | 132
    Asian - Central/South Asian Heritage | 20 | 19 | 39
    Asian - East Asian Heritage | 236 | 229 | 465
    Asian - Japanese Heritage | 1 | 2 | 3
    Asian - South East Asian Heritage | 81 | 81 | 162
    Native Hawaiian or Other Pacific Islander | 5 | 11 | 16
    White - Arabic/North African Heritage | 3 | 11 | 14
    White - White/Caucasian/European Heritage | 1126 | 1121 | 2247

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Par.) With Any Recurrence of the Initial Disease, Second Primary Cancer, Contralateral Breast Cancer, or Death (Disease-free Survival [DFS])
Description: DFS=interval between the date of randomization and the date of the first occurrence of an objective disease recurrence, a second primary cancer, or death from any cause. The date of the event is the earliest date of the occurrence of any of the following: local recurrence (LR) following mastectomy; LR in ipsilateral breast following lumpectomy; regional recurrence; distant recurrence; contralateral breast cancer, including ductal carcinoma in situ; other second primary cancer (excluding squamous or basal cell carcinoma of the skin, melanoma in situ, carcinoma in situ of the cervix, or lobular carcinoma in situ of the breast); death from any cause without a prior event. Par. who started additional anti-cancer adjuvant therapy prior to the recurrence of their disease were to be censored. Par. who did not withdraw from the study and did not experience a specified event or death were to be censored (follow-up ongoing) at the last visit date available at which progression was assessed.
Time Frame: From randomization until date of the first occurrence of an objective disease recurrence, a second primary cancer, or death from any cause (assessed up to 6 years; 1 year of treatment, 5 years of follow-up [median of 5.3 years for final analysis])
Population: Intent-to-Treat (ITT) Population: all randomized participants who received at least one dose of randomized treatment (lapatinib or placebo). Data for the end-of-study analysis (conducted in 2013) are reported.
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1571 | 1576
Participants
  Any recurrence or death | 252 | 290
  Censored, New Anti-cancer Agent/Radiotherapy | 1 | 1
  Censored, Follow-up Ended | 1318 | 1285
Statistical Analysis 1: Comparison: Lapatinib 1500 mg vs Placebo; Test type: Superiority or Other; p = 0.286, Log Rank — The p-value was calculated from a stratified log-rank test, stratifying for hormone receptor status, time since initial diagnosis, and lymph node involvement; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.77 to 1.08] — Estimate of the treatment hazard ratio (HR) was calcuated using the pike estimator

2. Secondary Outcome: Number of Participants Who Died (Overall Survival)
Description: Overall Survival (OS) is defined as the time from randomization until death from any cause. Data are presented as the number of participants who died. For participants who did not die, time to death was censored at the last date the participant was known to be alive.
Time Frame: From the date of randomization until death from any cause (assessed up to 6 years; 1 year of treatment and 5 years of follow-up [median of 5.3 years for final analysis])
Population: ITT Population. Data for the primary analysis (conducted in 2011) are reported.
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1571 | 1576
Participants
  Died | 115 | 126
  Censored, Follow-up Ended | 1456 | 1450

3. Secondary Outcome: Percentage of Participants With the Indicated Period of Recurrence-free Survival (Time to First Recurrence)
Description: Recurrence is defined as experiencing a recurrence of initial disease or contralateral breast cancer after randomization. Time to first recurrence is defined as the interval between the date of randomization and the date of the first occurrence of an objective disease recurrence or contralateral breast cancer. Time to first recurrence included the first occurrence at one of the following sites as an event: local recurrence following mastectomy; local recurrence in ipsilateral breast following lumpectomy; regional recurrence; distant recurrence; contralateral breast cancer, including ductal carcinoma in situ (DCIS).
Time Frame: From the date of randomization until the date of the first occurrence of an objective disease recurrence or contralateral breast cancer (assessed up to 6 years; 1 year of treatment and 5.3 years of follow-up [median of 5 years for final analysis])
Population: ITT Population. Data for the primary analysis (conducted in 2011) are reported.
Measure: Number; unit: Percentage of participants
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1571 | 1576
Percentage of participants
  6 Months | 1.3 | 2.8
  1Year | 3.7 | 5.4
  18 Months | 5.6 | 8.2
  2 Years | 7.7 | 9.9
  3 Years | 10.6 | 12.6
  4 Years | 13.3 | 15.8
  5 Years | NA — There was not sufficient follow-up to allow reasonable estimation of recurrence rates at time points beyond 5 years, when this analysis was carried out at the primary time point. | 24.9

4. Secondary Outcome: Percentage of Participants With the Indicated Period of Distant Recurrence-free Survival (Time to Distant Recurrence)
Description: Distant recurrence (metastatic disease) is defined as a tumor in any area of the body not including those defined as local or regional recurrence. Sites of distant recurrence include: skin, subcutaneous tissue, and lymph nodes (excluding those described for local and regional recurrence); bone marrow; skeletal; lungs and pleural; ascites and pleural effusions; liver and other viscera; and central nervous system (CNS). Time to distant recurrence is defined as the interval between the date of randomization and the date of the first occurrence of a distant recurrence.
Time Frame: From the date of randomization until the date of the first occurrence of a distant recurrence (assessed up to 6 years; 1 year of treatment and 5 years of follow-up [median of 5.3 years for final analysis])
Population: ITT Population. Data for the primary analysis (conducted in 2011) are reported.
Measure: Number; unit: Percentage of participants
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1571 | 1576
Percentage of participants
  6 Months | 0.9 | 1.9
  1Year | 2.9 | 3.8
  18 Months | 4.3 | 6.0
  2 Years | 5.9 | 7.2
  3 Years | 8.1 | 9.1
  4 Years | 9.3 | 11.1
  5 Years | NA — There was not sufficient follow-up to allow reasonable estimation of recurrence rates at time points beyond 5 years, when this analysis was carried out at the primary time point. | 14.2

5. Secondary Outcome: Time to Central Nervous System (CNS) Recurrence
Description: Time to CNS recurrence is defined as the interval between the date of randomization and the date of the occurrence of a CNS recurrence if noted as part of the participant's first recurrence. Time to CNS recurrence was not calculated; data are presented as the number of participants with CNS recurrence in the subsequent outcome measure table.
Time Frame: From the date of randomization until the date of the first occurrence of a CNS recurrence (assessed up to 6 years [1 year of treatment and 5 years of follow-up; median of 5.3 years for final analysis])
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With CNS Recurrence
Description: The number of participants experiencing a CNS recurrence was summarized.
Time Frame: as for outcome 5
Population: ITT Population. Data for the end-of-study analysis (conducted in 2013) are reported.
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1571 | 1576
Participants | 15 | 21

7. Secondary Outcome: Modified Disease-free Survival (MDFS)
Description: Modified disease recurrence=interval between the date of randomization and the date of the first occurrence of an objective disease recurrence, contralateral breast cancer, or death from any cause. The date of the event=the earliest date of the occurrence of any of the following events: local recurrence following mastectomy; local recurrence in ipsilateral breast following lumpectomy; regional recurrence; distant recurrence; contralateral breast cancer, including DCIS; death from any cause without a prior event. MDFS was not calculated; data are presented as the number of participants with any recurrence of the initial disease, contralateral breast cancer, or death (disease-free survival) in the subsequent outcome measure table.
Time Frame: From the date of randomization until the date of the first occurrence of an objective disease recurrence, contralateral breast cancer, or death from any cause (assessed up to 6 years)
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Any Recurrence of the Initial Disease, Contralateral Breast Cancer, or Death (Disease-free Survival [DFS])
Description: DFS=interval between the date of randomization and the date of the first occurrence of an objective disease recurrence, a second primary cancer, or death from any cause. The date of the event is the earliest date of the occurrence of any of the following: local recurrence (LR) following mastectomy; LR in ipsilateral breast following lumpectomy; regional recurrence; distant recurrence and contralateral breast cancer, including ductal carcinoma in situ; or death from any cause without a prior event. Participants who started additional anti-cancer adjuvant therapy prior to the recurrence of their disease were to be censored. Participants who did not withdraw from the study and did not experience a specified event or death were to be censored (follow-up ongoing) at the last visit date available at which progression was assessed.
Time Frame: as for outcome 7
Population: ITT Population. Data for the end-of-study analysis (conducted in 2013) are reported.
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1571 | 1576
Participants | 184 | 231

9. Secondary Outcome: Change From Baseline in Short Form-36 Version 2 (SF-36 v2) Scores for the Physical Component Summary (PCS)
Description: The SF-36 v2 is a self-administered, health-related quality of life (QoL) metric. It is a 36-item questionnaire designed to measure 8 domains of functional health status and well-being: physical functioning, role-physical, bodily pain, general health perceptions, vitality, social functioning, role-emotional, and mental health. Each domain is scored from 0 (poorer health) to 100 (better health).The PCS score is a summary score representing overall physical health, which is derived from the 8 domain scores. As with each domain score, the PCS score ranges from 0 to 100; higher scores represent better health. Change from Baseline was calculated as the post-Baseline score minus the Baseline score. Missing post-Baseline data were imputed using the last observation carried forward (LOCF) method. The scores were analyzed using an analysis of covariance (ANCOVA) model, adjusting for Baseline sub-scale score, treatment, and country. Positive changes from Baseline indicate improvement.
Time Frame: Baseline, Month 6, Month 12, and every 6 months after discontinuation of study treatment for 24 months (up to a maximum of 3 study years)
Population: ITT Population (primary analysis [conducted in 2011]). Only those participants available (represented as n=X, X in the category titles) at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1092 | 1283
Scores on a scale
  Month 6, n=1092, 1283 | -0.78 (0.217) | -0.44 (0.211)
  Month 12, n=1007, 1204 | -0.84 (0.251) | -0.54 (0.242)
  Follow-up, Month 6, n= 983, 1074 | -0.53 (0.287) | -0.87 (0.281)
  Follow-up, Month 12, n= 940, 988 | -0.88 (0.290) | -0.82 (0.289)
  Follow-up, Month 18, n=834, 889 | -0.61 (0.350) | -0.89 (0.346)
  Follow-up, Month 24, n=807, 824 | -0.99 (0.412) | -0.66 (0.417)
  Early inv. product discontinuation, n=289, 120 | -4.39 (0.712) | -4.00 (0.886)

10. Secondary Outcome: Change From Baseline in SF-36 v2 Scores for the Mental Component Summary (MCS)
Description: The SF-36 v2 is a self-administered, health-related quality of life (QoL) metric. It is a 36-item questionnaire designed to measure 8 domains of functional health status and well-being: physical functioning, role-physical, bodily pain, general health perceptions, vitality, social functioning, role-emotional, and mental health. Each domain is scored from 0 (poorer health) to 100 (better health).The MCS score is a summary score representing overall mental health, which is derived from the 8 domain scores. As with each domain score, the MCS score ranges from 0 to 100; higher scores represent better health. Change from Baseline was calculated as the post-Baseline score minus the Baseline score. Missing post-Baseline data were imputed using the LOCF method. The scores were analyzed using an ANCOVA model adjusting for Baseline sub-scale score, treatment, and country. Positive changes from Baseline indicate improvement.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1092 | 1283
Scores on a scale
  Month 6, n=1092, 1283 | -2.34 (0.306) | -1.74 (0.297)
  Month 12, n=1007, 1204 | -2.74 (0.332) | -2.29 (0.322)
  Follw-up, Month 6, n=983, 1074 | -2.22 (0.368) | -1.87 (0.361)
  Follow-up, Month 12, n= 940, 988 | -3.08 (0.393) | -2.76 (0.392)
  Follow-up, Month 18, n=834, 889 | -2.38 (0.480) | -2.08 (0.475)
  Follow-up, Month 24, n=807, 824 | -2.78 (0.547) | -3.05 (0.554)
  Early inv. product discontinuation, n=289, 120 | -6.65 (0.985) | -8.11 (1.221)

11. Secondary Outcome: Change From Baseline in the SF-36 v2 Domain Scores for Physical Functioning (PF), Role-Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role-Emotional (RE), and Mental Health (MH)
Description: The SF-36 v2 is a self-administered, health-related quality of life (QoL) metric. It is a 36-item questionnaire designed to measure 8 domains of functional health status and well-being: physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH) perceptions, vitality (VT), social functioning (SF), role-emotional (RE), and mental health (MH). Each domain is scored from 0 (poorer health) to 100 (better health); higher scores represent better health. Change from Baseline was calculated as the post-Baseline score minus the Baseline score. Missing post-Baseline data were imputed using the LOCF method. The scores were analyzed using an ANCOVA model, adjusting for Baseline sub-scale score, treatment, and country. Positive changes from Baseline indicate improvement.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1132 | 1345
Scores on a scale
  PF, Month 6, n=1132, 1345 | -0.52 (0.235) | -0.65 (0.227)
  PF, Month 12, n=1025, 1234 | -0.59 (0.269) | -0.91 (0.260)
  PF, Follow-up, Month 6, n=997, 1097 | -0.45 (0.296) | -0.81 (0.289)
  PF, Follow-up, Month 12, n=955, 1013 | -1.11 (0.317) | -1.40 (0.316)
  PF, Follow-up, Month 18, n=851, 913 | -0.80 (0.363) | -1.10 (0.358)
  PF, Follow-up, Month 24, n=818, 845 | -1.06 (0.438) | -1.17 (0.442)
  PF, Early inv. Product discontinuation, n=304, 128 | -4.30 (0.755) | -4.43 (0.928)
  RP, Month 6, n=1130, 1335 | -1.37 (0.276) | -0.87 (0.267)
  RP, Month 12, n=1023, 1230 | -1.52 (0.303) | -0.83 (0.293)
  RP, Follow-up, Month 6, n=997, 1094 | -1.14 (0.328) | -1.45 (0.322)
  RP, Follow-up, Month 12, n=955, 1009 | -1.78 (0.344) | -1.47 (0.343)
  RP, Follow-up, Month 18, n=851, 909 | -1.72 (0.410) | -1.68 (0.405)
  RP, Follow-up, Month 24, n=818, 842 | -1.77 (0.486) | -1.54 (0.491)
  RP, Early inv. product discontinuation, n=303, 127 | -6.96 (0.882) | -7.09 (1.087)
  BP, Month 6, n=1130, 1331 | -1.58 (0.304) | -1.31 (0.295)
  BP, Month 12, n=1024, 1229 | -1.75 (0.338) | -1.62 (0.326)
  BP, Follow-up, Month 6, n=995, 1094 | -1.13 (0.376) | -1.35 (0.368)
  BP, Follow-up, Month 12, n=954, 1007 | -1.06 (0.383) | -1.19 (0.382)
  BP, Follow-up, Month 18, n=847, 909 | -0.69 (0.461) | -1.07 (0.455)
  BP, Follow-up, Month 24, n=817, 840 | -1.69 (0.547) | -1.41 (0.553)
  BP, Early inv. product discontinuation, n=302, 126 | -4.92 (0.950) | -4.97 (1.164)
  GH, Month 6, n=1124, 1319 | -1.01 (0.244) | -0.34 (0.236)
  GH, Month 12, n=1020, 1221 | -1.33 (0.275) | -0.70 (0.266)
  GH, Follow-up, Month 6, n=994, 1085 | -1.25 (0.314) | -1.34 (0.308)
  GH, Follow-up, Month 12, n=951, 1002 | -1.93 (0.330) | -1.48 (0.329)
  GH, Follow-up, Month 18, n=844, 902 | -1.28 (0.397) | -1.28 (0.392)
  GH, Follow-up, Month 24, n=813, 835 | -1.29 (0.471) | -1.02 (0.476)
  GH, Early inv. product discontinuation, n=299, 124 | -5.12 (0.775) | -6.30 (0.965)
  VT, Month 6, n=1126, 1332 | -2.30 (0.283) | -1.83 (0.274)
  VT, Month 12, n=1022, 1225 | -2.49 (0.309) | -1.88 (0.299)
  VT, Follow-up, Month 6, n=993, 1090 | -1.55 (0.335) | -1.61 (0.328)
  VT, Follow-up, Month 12, n=953, 1006 | -2.45 (0.355) | -2.01 (0.354)
  VT, Follow-up, Month 18, n=848, 906 | -1.53 (0.426) | -1.25 (0.421)
  VT, Follow-up, Month 24, n=817, 837 | -2.03 (0.501) | -1.96 (0.507)
  VT, Early inv. product discontinuation, n=303, 125 | -5.54 (0.867) | -5.78 (1.067)
  SF, Month 6, n=1138, 1347 | -2.34 (0.299) | -1.42 (0.289)
  SF, Month 12, n=1025, 1234 | -2.63 (0.333) | -2.05 (0.322)
  SF, Follow-up, Month 6, n=997, 1098 | -1.80 (0.371) | -1.51 (0.363)
  SF, Follow-up, Month 12, n=957, 1011 | -2.47 (0.383) | -2.17 (0.382)
  SF, Follow-up, Month 18, n=850, 912 | -1.96 (0.462) | -2.01 (0.456)
  SF, Follow-up, Month 24, n=819, 843 | -2.94 (0.526) | -2.75 (0.532)
  SF, Early inv. product discontinuation, n=305, 127 | -7.05 (1.017) | -7.94 (1.247)
  RE, Month 6, n=1124, 1328 | -1.80 (0.335) | -1.69 (0.325)
  RE, Month 12, n=1023, 1226 | -1.99 (0.357) | -1.99 (0.345)
  RE, Follow-up, Month 6, n=996, 1091 | -1.87 (0.393) | -1.88 (0.385)
  RE, Follow-up, Month 12, n=955, 1004 | -2.88 (0.425) | -2.72 (0.425)
  RE, Follow-up,Month 18, n=851, 905 | -2.47 (0.509) | -2.50 (0.503)
  RE, Follow-up,Month 24, n=818, 839 | -2.75 (0.582) | -2.95 (0.589)
  RE, Early inv. product discontinuation, n=303, 126 | -6.85 (1.020) | -8.00 (1.258)
  MH, Month 6, n=1124, 1332 | -1.96 (0.303) | -1.46 (0.293)
  MH, Month 12, n=1021, 1225 | -2.38 (0.333) | -2.11 (0.322)
  MH, Follow-up, Month 6, n=993, 1090 | -1.92 (0.367) | -1.70 (0.360)
  MH, Follow-up, Month 12, n=953, 1006 | -2.47 (0.390) | -2.47 (0.389)
  MH, Follow-up, Month 18, n=848, 906 | -1.91 (0.469) | -1.58 (0.464)
  MH, Follow-up, Month 24, n=817, 837 | -2.16 (0.545) | -2.54 (0.552)
  MH, Early inv. product discontinuation, n=303, 125 | -5.96 (0.964) | -7.87 (1.187)

12. Secondary Outcome: Number of Participants With Hematology Values Outside the Reference Range for the Indicated Parameters
Description: The hematology parameters assessed were: basophils (Bs) in giga (10^9) per liter (GI/L) and in percentage (%), eosinophils (Eo) in GI/L and %, hematocrit, hemoglobin, lymphocytes (Lmph) in GI/L and %, monocytes (Mono) in GI/L and %, platelet count, Red Blood Cell (RBC) count, total neutrophil count (TNC) in GI/L and %, and White Blood Cell (WBC) count. The Baseline (BL) value is the last available pre-treatment result recorded. "Any post-Baseline value" was based on results recorded at any scheduled or unscheduled post-Baseline visits. The prevalence of values lying outside the reference (ref.) range (high or low) is presented for BL and "any post-Baseline" (APBL) visit. Two participants were randomized to placebo but received lapatinib; therefore, they are included in the lapatinib treatment arm. Data for the primary analysis (conducted in 2011) are reported.
Time Frame: At Baseline and every 3 months thereafter up to Month 12/Early Withdrawal Visit
Population: Safety Population (SP): all randomized participants (par.) who received >=1 dose of randomized treatment. Only those par. available (n=X, X in the category titles) at the specified time points were analyzed. Different par. may have been analyzed for different parameters, so the overall number of par. analyzed reflects everyone in the SP.
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1573 | 1574
Participants
  Bs (GI/L), BL, ref. range high, n=1555, 1563 | 0 | 1
  Bs (GI/L), BL, ref. range low, n=1555, 1563 | 0 | 0
  Bs (GI/L), APBL, ref. range high, n=1466, 1537 | 7 | 7
  Bs (GI/L), APBL, ref. range low, n=1466, 1537 | 7 | 2
  Eo (GI/L), BL, ref. range high, n=1557, 1562 | 34 | 35
  Eo (GI/L), BL, ref. range low, n=1557, 1562 | 242 | 184
  Eo (GI/L), APBL, ref. range high, n=1466, 1537 | 84 | 75
  Eo (GI/L), APBL, ref. range low, n=1466, 1537 | 322 | 370
  Hematocrit, BL, ref. range high, n=1560, 1563 | 20 | 30
  Hematocrit, BL, ref. range low, n=1560, 1563 | 72 | 96
  Hematocrit, APBL, ref. range high, n=1474, 1538 | 46 | 65
  Hematocrit, APBL, ref. range low, n=1474, 1538 | 196 | 145
  Hemoglobin, BL, ref. range high, n=1560, 1563 | 8 | 16
  Hemoglobin, BL, ref. range low, n=1560, 1563 | 148 | 160
  Hemoglobin, APBL, ref. range high, n=1474, 1538 | 32 | 34
  Hemoglobin, APBL, ref. range low, n=1474, 1538 | 295 | 212
  Lmph (GI/L), BL, ref. range high, n=1557, 1562 | 5 | 1
  Lmph (GI/L), BL, ref. range low, n=1557, 1562 | 80 | 89
  Lmph (GI/L), APBL, ref. range high, n=1468, 1538 | 12 | 11
  Lmph (GI/L), APBL, ref. range low, n=1468, 1538 | 106 | 100
  Mono (GI/L), BL, ref. range high, n=1557, 1562 | 2 | 4
  Mono (GI/L), BL, ref. range low, n=1557, 1562 | 236 | 239
  Mono (GI/L), APBL, ref. range high, n=1466, 1538 | 7 | 7
  Mono (GI/L), APBL, ref. range low, n=1466, 1538 | 425 | 431
  Platelet count, BL, ref. range high, n=1553, 1559 | 34 | 33
  Platelet count, BL, ref. range low, n=1553, 1559 | 21 | 15
  Platelet count, APBL, ref. range high, n=1473, 153 | 95 | 56
  Platelet count, APBL, ref. range low, n=1473, 1538 | 40 | 37
  RBC count, BL, ref. range high, n=1559, 1563 | 10 | 18
  RBC count, BL, ref. range low, n=1559, 1563 | 144 | 148
  RBC count, APBL, ref. range high, n=1474, 1538 | 25 | 36
  RBC count, APBL, ref. range low, n=1474, 1538 | 270 | 207
  TNC (GI/L), BL, ref. range high, n=1557, 1563 | 17 | 15
  TNC (GI/L), BL, ref. range low, n=1557, 1563 | 47 | 41
  TNC (GI/L), APBL, ref. range high, n=1469, 1538 | 38 | 53
  TNC (GI/L), APBL, ref. range low, n=1469, 1538 | 115 | 161
  WBC count, BL, ref. range high, n=1559, 1563 | 18 | 14
  WBC count, BL, ref. range low, n=1559, 1563 | 142 | 104
  WBC count, APBL, ref. range high, n=1471, 1537 | 42 | 57
  WBC count, APBL, ref. range low, n=1471, 1537 | 191 | 198
  Bs (%), BL, ref. range high, n=64, 55 | 8 | 4
  Bs (%), BL, ref. range low, n=64, 55 | 1 | 0
  Bs (%), APBL, ref. range high, n=131, 131 | 17 | 18
  Bs (%), APBL, ref. range low, n=131, 131 | 4 | 1
  Eo (%), BL, ref. range high, n=65, 55 | 7 | 9
  Eo (%), BL, ref. range low, n=65, 55 | 2 | 1
  Eo (%), APBL, ref. range high, n=135, 132 | 16 | 20
  Eo (%), APBL, ref. range low, n=135, 132 | 9 | 4
  Lmph (%), BL, ref. range high, n=68, 57 | 4 | 3
  Lmph (%), BL, ref. range low, n=68, 57 | 10 | 10
  Lmph (%), APBL, ref. range high, n=152, 143 | 14 | 18
  Lmph (%), APBL, ref. range low, n=152, 143 | 19 | 16
  Mono (%), BL, ref. range high, n=67, 54 | 13 | 11
  Mono (%), BL, ref. range low, n=67, 54 | 0 | 0
  Mono (%), APBL, ref. range high, n=137, 139 | 28 | 11
  Mono (%), APBL, ref. range low, n=137, 139 | 6 | 4
  TNC (%), BL, ref. range high, n=68, 58 | 7 | 2
  TNC (%), BL, ref. range low, n=68, 58 | 5 | 4
  TNC (%), APBL, ref. range high, n=150, 145 | 9 | 10
  TNC (%), APBL, ref. range low, n=150, 145 | 19 | 12

13. Secondary Outcome: Number of Participants With Clinical Chemistry Values Outside the Reference Range for the Indicated Parameters
Description: The clinical chemistry parameters assessed were: alanine amino transferase (ALT), albumin, alkaline phosphatase (ALP), aspartate amino transferase (AST), bicarbonate, blood urea nitrogen (BUN), bone alkaline phosphatase (Bone ALP), calcium, chloride, creatinine, creatinine clearance (Cr. Clearance), creatinine clearance estimated (Cr. Clrnc. est.), glucose, potassium, sodium, total bilirubin (Total Bln), total protein, urea, and uric acid. The Baseline (BL) value is the last available pre-treatment result recorded. "Any post-Baseline" value was based on results recorded at scheduled or unscheduled post-Baseline visits. The prevalence of values lying outside the reference (ref.) range (high or low) was presented for BL and "any post-Baseline" (APBL) visit. Two participants were randomized to placebo but received lapatinib; therefore, they are included in the lapatinib treatment arm.
Time Frame: At Baseline and every 6 weeks thereafter up to Month 12/Early Withdrawal Visit
Population: Safety Population (primary analysis [conducted in 2011]). Only those participants available (represented as n=X, X in the category titles) at the specified time points were analyzed. Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the Safety Population.
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1573 | 1574
Participants
  ALT, BL, ref. range high, n=1569, 1569 | 55 | 78
  ALT, BL, ref. range low, n=1569, 1569 | 1 | 1
  ALT, APBL, ref. range high, n=1478, 1542 | 271 | 141
  ALT, APBL, ref. range low, n=1478, 1542 | 3 | 5
  Albumin, BL, ref. range high, n=1568, 1568 | 36 | 41
  Albumin, BL, ref. range low, n=1568, 1568 | 0 | 0
  Albumin, APBL, ref. range high, n=1475, 1542 | 51 | 70
  Albumin, APBL, ref. range low, n=1475, 1542 | 11 | 8
  ALP, BL, ref. range high, n=1569, 1569 | 68 | 66
  ALP, BL, ref. range low, n=1569, 1569 | 0 | 0
  ALP, APBL, ref. range high, n=1477, 1542 | 213 | 155
  ALP, APBL, ref. range low, n=1477, 1542 | 4 | 5
  AST, BL, ref. range high, n=1569, 1565 | 49 | 59
  AST, BL, ref. range low, n=1569, 1565 | 0 | 0
  AST, APBL, ref. range high, n=1478, 1541 | 260 | 139
  AST, APBL, ref. range low, n=1478, 1541 | 0 | 3
  Bicarbonate, BL, ref. range high, n=36, 33 | 0 | 3
  Bicarbonate, BL, ref. range low, n=36, 33 | 4 | 3
  Bicarbonate, APBL, ref. range high, n=60, 71 | 3 | 2
  Bicarbonate, APBL, ref. range low, n=60, 71 | 4 | 9
  BUN, BL, ref. range high, n=63, 56 | 8 | 4
  BUN, BL, ref. range low, n=63, 56 | 0 | 0
  BUN, APBL, ref. range high, n=161, 155 | 15 | 17
  BUN, APBL, ref. range low, n=161, 155 | 6 | 4
  Bone ALP, BL, ref. range high, n=230, 219 | 0 | 0
  Bone ALP, BL, ref. range low, n=230, 219 | 0 | 0
  Bone ALP, APBL, ref. range high, n=188, 160 | 0 | 0
  Bone ALP, APBL, ref. range low, n=188, 160 | 0 | 0
  Calcium, BL, ref. range high, n=1568, 1565 | 17 | 36
  Calcium, BL, ref. range low, n=1568, 1565 | 16 | 14
  Calcium, APBL, ref. range high, n=1476, 1542 | 56 | 84
  Calcium, APBL, ref. range low, n=1476, 1542 | 66 | 79
  Chloride, BL, ref. range high, n=52, 46 | 2 | 2
  Chloride, BL, ref. range low, n=52, 46 | 0 | 1
  Chloride, APBL, ref. range high, n=102, 108 | 10 | 5
  Chloride, APBL, ref. range low, n=102, 108 | 2 | 5
  Creatinine, BL, ref. range high, n=1569, 1569 | 5 | 4
  Creatinine, BL, ref. range low, n=1569, 1569 | 7 | 8
  Creatinine, APBL, ref. range high, n=1479, 1542 | 16 | 13
  Creatinine, APBL, ref. range low, n=1479, 1542 | 22 | 27
  Cr. Clearance, BL, ref. range high, n=4, 9 | 2 | 2
  Cr. Clearance, BL, ref. range low, n=4, 9 | 1 | 0
  Cr. Clearance, APBL, ref. range high, n=11, 10 | 0 | 1
  Cr. Clearance, APBL, ref. range low, n=11, 10 | 2 | 2
  Cr. Clrnc. est., BL, ref. range high, n=373, 388 | 0 | 0
  Cr. Clrnc. est., BL, ref. range low, n=373, 388 | 0 | 0
  Cr. Clrnc. est., APBL, ref. range high, n=380, 418 | 0 | 0
  Cr. Clrnc. est., APBL, ref. range low, n=380, 418 | 0 | 0
  Glucose, BL, ref. range high, n=1566, 1569 | 170 | 143
  Glucose, BL, ref. range low, n=1566, 1569 | 31 | 32
  Glucose, APBL, ref. range high, n=1475, 1541 | 245 | 329
  Glucose, APBL, ref. range low, n=1475, 1541 | 94 | 94
  Potassium, BL, ref. range high, n=1567, 1565 | 13 | 13
  Potassium, BL, ref. range low, n=1567, 1565 | 21 | 11
  Potassium, APBL, ref. range high, n=1476, 1542 | 28 | 54
  Potassium, APBL, ref. range low, n=1476, 1542 | 54 | 44
  Sodium, BL, ref. range high, n=1568, 1568 | 9 | 4
  Sodium, BL, ref. range low, n=1568, 1568 | 7 | 9
  Sodium, APBL, ref. range high, n=1477, 1542 | 29 | 27
  Sodium, APBL, ref. range low, n=1477, 1542 | 24 | 30
  Total Bln., BL, ref. range high, n=1569, 1569 | 14 | 19
  Total Bln., BL, ref. range low, n=1569, 1569 | 1 | 0
  Total Bln., APBL, ref. range high, n=1478, 1542 | 152 | 46
  Total Bln., APBL, ref. range low, n=1478, 1542 | 4 | 3
  Total Protein, BL, ref. range high, n=1566, 1568 | 3 | 9
  Total Protein, BL, ref. range low, n=1566, 1568 | 4 | 1
  Total Protein, APBL, ref. range high, n=1476, 1542 | 27 | 38
  Total Protein, APBL, ref. range low, n=1476, 1542 | 11 | 13
  Urea, BL, ref. range high, n=1560, 1566 | 18 | 19
  Urea, BL, ref. range low, n=1560, 1566 | 17 | 24
  Urea, APBL, ref. range high, n=1465, 1535 | 35 | 48
  Urea, APBL, ref. range low, n=1465, 1535 | 45 | 48
  Uric acid, BL, ref. range high, n=37, 26 | 7 | 5
  Uric acid, BL, ref. range low, n=37, 26 | 0 | 1
  Uric acid, APBL, ref. range high, n=73, 76 | 10 | 12
  Uric acid, APBL, ref. range low, n=73, 76 | 3 | 4

14. Secondary Outcome: Number of Participants With Non-laboratory Toxicities of the Indicated Toxicity Grades
Description: Non-laboratory toxicities are defined as adverse events (AEs). The number of partcipants with any treatment-emergent AE of the indicated toxicity grade are summarized. Toxicity grading was according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0 as follows: Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life threatening; Grade 5=death. The events that were not given a toxicity grade are categorized as "Not Applicable."
Time Frame: From the first dose of study treatment up to 12 months
Population: Safety Population. Two participants were randomized to placebo but received lapatinib; therefore, they are included in the lapatinib treatment arm. Data for the primary analysis (conducted in 2011) are reported.
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1573 | 1574
Participants
  Grade 1 | 414 | 558
  Grade 2 | 674 | 505
  Grade 3 | 333 | 104
  Grade 4 | 21 | 15
  Grade 5 | 3 | 3
  Not Applicable | 5 | 8

15. Secondary Outcome: Number of Participants Experiencing Primary or Secondary Cardiac Events
Description: A cardiac event is classified as a primary cardiac endpoint (PCE) or a secondary cardiac endpoint (SCE). PCE is defined as: cardiac death (cardiac death due to heart failure, myocardial infarction, or arrhythmia;or probable cardiac death defined as sudden, unexpected death within 24 hours of a definite or probable cardiac event); severe symptomatic congestive heart failure (CHF) (as per New York Heart Association [NYHA] Class III or IV and an absolute decrease in left ventricular ejection fraction [LVEF] of more than 10 percentage points from Baseline and to a left ventricular ejection fraction [LVEF] value below 50%). SCE is defined as asymptomatic or mildly symptomatic cardiac events (NYHA Class I or II) and a significant decrease in LVEF, defined as an absolute decrease in LVEF of more than 10 percentage points from Baseline and to an LVEF value below 50%.
Time Frame: From the date of randomization up to 12 months
Population: Safety Population (SP). Two participants were randomized to placebo but received lapatinib; therefore, they are included in the lapatinib treatment arm. Data for the primary analysis (conducted in 2011) are reported.
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1573 | 1574
Participants
  PCE, Cardiac death | 0 | 1
  PCE, Severe symptomatic CHF | 2 | 3
  SCE | 6 | 6

16. Secondary Outcome: Number of Participants With the Indicated Electrocardiogram (ECG) Findings
Description: 12-lead ECG measurements were taken at Screening and at study conclusion/withdrawal. The number of participants with normal, abnormal clinically significant (CS), and abnormal not clinically significant (NCS) ECG findings, as classified by the investigator, were summarized. Participants with missing values were categorized as missing. Data for the primary analysis (conducted in 2011) are reported.
Time Frame: Screening and Month 12/Early Withdrawal Visit
Population: SP. Only those participants (par.) available at the specified time points were analyzed. Two par. were randomized to placebo but received lapatinib; therefore, they are included in the lapatinib treatment arm.
Measure: Number; unit: Participants
Arm/Group | Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 1543 | 1549
Participants
  Screening, normal, n=1543, 1549 | 1203 | 1197
  Screening, abnormal CS, n=1543, 1549 | 0 | 1
  Screening, abnormal NCS, n=1543, 1549 | 339 | 351
  Screening, missing, n=1543, 1549 | 1 | 0
  Conclusion/ Withdrawal, normal, n=1243, 1306 | 960 | 979
  Conclusion/ Withdrawal, abnormal CS, n=1243, 1306 | 5 | 3
  Conclusion/ Withdrawal, abnormal NCS, n=1243, 1306 | 276 | 323
  Conclusion/ Withdrawal, missing, n=1243, 1306 | 2 | 1

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (AEs): collected from start of treatment until up to 5 days after the last dose of study treatment (up to 12 months). SAEs: collected up to any time during the follow-up period post discontinuation of study drug (up to 6 years).
Description: Non-serious AEs and SAEs were collected in members of the Safety Population, comprised of all randomized participants who received at least one dose of randomized treatment. Two participants were randomized to placebo but received lapatinib; therefore, they are included in the lapatinib treatment arm.
Arm/Group | Lapatinib 1500 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 99/1573 | 78/1574
Other Adverse Events (participants affected / at risk) | 1443/1573 | 1175/1574
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1500 mg (N=1573) | Placebo (N=1574)
Erysipelas (Infections and infestations) | 8 | 0
Cellulitis (Infections and infestations) | 5 | 0
Pneumonia (Infections and infestations) | 3 | 2
Appendicitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 2 | 0
Abscess (Infections and infestations) | 1 | 0
Breast abscess (Infections and infestations) | 0 | 1
Breast cellulitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Implant site cellulitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Contralataral breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinaom metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Enteritis (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Infections and infestations) | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 3 | 1
Cardiac failure (Cardiac disorders) | 0 | 3
Myocardial infarction (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ejection fraction decreased (Investigations) | 5 | 6
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin abnormal (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road tracffic accident (Injury, poisoning and procedural complications) | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Ovarian enlargement (Reproductive system and breast disorders) | 0 | 1
Asthenia (General disorders) | 0 | 2
Death (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Capillary leak syndrome (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Thyroiditis subacute (Endocrine disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib 1500 mg (N=1573) | Placebo (N=1574)
Diarrhoea (Gastrointestinal disorders) | 955 | 256
Rash (Skin and subcutaneous tissue disorders) | 922 | 243
Nausea (Gastrointestinal disorders) | 279 | 179
Fatigue (General disorders) | 251 | 202
Headache (Nervous system disorders) | 140 | 185
Dry skin (Skin and subcutaneous tissue disorders) | 220 | 45
Arthralgia (Musculoskeletal and connective tissue disorders) | 69 | 113
Pruritus (Skin and subcutaneous tissue disorders) | 130 | 49
Cough (Respiratory, thoracic and mediastinal disorders) | 75 | 103
Vomiting (Gastrointestinal disorders) | 104 | 71
Dyspepsia (Gastrointestinal disorders) | 106 | 57
Abdominal pain (Gastrointestinal disorders) | 105 | 56
Alopecia (Skin and subcutaneous tissue disorders) | 135 | 25
Paronychia (Infections and infestations) | 154 | 5
Nail disorder (Skin and subcutaneous tissue disorders) | 131 | 16
Decreased appetite (Metabolism and nutrition disorders) | 99 | 36
Stomatitis (Eye disorders) | 98 | 30
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 118 | 8
Skin fissures (Skin and subcutaneous tissue disorders) | 83 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.